CLINICAL TRIAL: NCT06434090
Title: Liposomal Irinotecan Plus Bevacizumab in Irinotecan-refractory Metastatic Colorectal Cancer:a Multicenter, Phase I/II Trial.
Brief Title: Liposomal Irinotecan Plus Bevacizumab in Irinotecan-refractory Metastatic Colorectal Cancer
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yanhong Deng, Director of Medical Oncology, Clinical Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSPC-DEY-CRC-K06
Record Dates: First submitted 2024-05-23; First posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Colorectal Cancer
Keywords: Liposomal irinotecan; bevacizumab
MeSH Terms: conditions — Colorectal Neoplasms | interventions — irinotecan sucrosofate; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Liposomal irinotecan plus bevacizumab (Experimental): Patients received Liposomal irinotecan (a '3+3' design was adopted in the experimental arm, with 3 dose levels of 70mg/m2, 80mg/m2, and 90mg/m2 for dose exploration) every 2 weeks (Q2W).
  bevacizumab, 5mg/m2, every 2 weeks The two-drug combination therapy was continued every 2 weeks in a cycle until patients developed disease progression or met other criteria for termination of study treatment specified in the protocol.
  Interventions: Drug: Liposomal irinotecan; Drug: Bevacizumab

INTERVENTIONS:
Drug: Liposomal irinotecan — Liposomal irinotecan will be given biweekly at a dose from 70mg/m2 to 90mg/m2.
Drug: Bevacizumab — bevacizumab will be given biweekly at a dose of 5mg/m2
  Other Names: avastin

SUMMARY:
To evaluate the efficacy and safety of liposomal irinotecan plus bevacizumab in irinotecan-refractory metastatic colorectal cancer

DETAILED DESCRIPTION:
The standard treatment regimen based on irinotecan with or without bevacizumab is commonly used in metastatic colorectal cancer. With administration of traditional irinotecan, the parent drug and active metabolite SN-38 exist in the form of active lactone and carboxylate, and the lactone ring structure is unstable in neutral and alkaline solutions. In physiological pH conditions, the active lactone rapidly hydrolyzes to the inactive carboxylate, thereby reducing the efficacy, so there is certain limitation in clinical application.

Liposomes Irinotecan load the active substance irinotecan into liposomes, so that it can be slowly released in the body and achieve the effect of reducing toxicity and increasing efficacy.After being rationally designed, irinotecan liposomes can also take advantage of the high permeability and retention effect (EPR) to specifically target the tumor area, increase the amount of drug taken up by cancer cells, reduce the dosage, improve efficacy, and reduce side effects.

We are currently conducting an Phase I/II study in mCRC patients who have previously received irinotecan. After determining the maximum tolerable dose (MTD) of irinotecan liposomes in the combined regimen of irinotecan liposomes and bevacizumab, we will further explore the safety and initial efficacy of irinotecan liposomes combined with bevacizumab.

ELIGIBILITY:
Inclusion Criteria:

1. Age: ≥18 years old；
2. Histopathologically and/or cytologically confirmed unresectable metastatic colorectal adenocarcinoma；
3. Previous treatment with irinotecan , and have progression of disease during treatment or within three months thereafter；
4. At least one measurable lesion (according to RECIST v1.1)；
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 ~ 1；
6. The expected survival time ≥3 months；
7. Adequate bone marrow function : no blood transfusion and/or use of increasing leukocyte drugs (excluding oral medication) within 14 days prior to enrollment Absolute neutrophil count (ANC) ≥1.5×109/L Platelet count ≥100×109/L Hemoglobin (Hgb) ≥90 g/L；
8. Adequate hepatic function as evidenced by:

Total bilirubin ≤1.5 × upper limit of normal (ULN), Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 × ULN, ≤5 × ULN if liver metastases are present.

Serum albumin ≥30 g/L； (9Adequate renal function as evidenced by: serum creatinine (Cr) ≤1.5 × ULN or creatinine clearance ≥60 mL/min. proteinuria<2+（those with proteinuria ≥2+ at baseline had to demonstrate ≤1 g protein per 24 hours）； (10)Coagulation function: International normalised ratio (INR) ≤1.5, activated partial thromboplastin time (APTT) ≤1.5 × ULN； (11)Agree and be able to comply with the plan during the study period. Provide written informed consent before entering the study screening；

Exclusion Criteria:

1. Any other malignancy within 5 years, with the exception of cured in-situ carcinoma or basal cell carcinoma etc；
2. Patients with the primary lesion located in the left colon and RAS/BRAF wild-type who did not use cetuximab on the first-line；
3. Patients with high microsatellite instability (MSI-H) or mismatch repair deficiency (dMMR)；
4. Massive pleural effusion or ascites requiring intervention；
5. Active, uncontrolled bacterial, viral, or fungal infections that require systemic treatment；
6. Active HIV infection；
7. Combined with uncontrollable systemic diseases within 6 months before the first administration；
8. Presence of severe gastrointestinal disease；
9. History of major surgery (such as laparotomy, thoracotomy or intestinal resection) within 28 days before the first administration,or plan to undergo major surgery during the study period；
10. Presence of interstitial pneumonia or pulmonary fibrosis；
11. History of allergy or hypersensitivity to drug or any of their excipients；
12. History of pulmonary hemorrhage/hemoptysis ≥Grade 2 (defined as bright red blood of at least 2.5mL) within one month before the first administration；
13. Presence of arterial embolism, severe bleeding (excluding bleeding caused by surgery) or tendency for existing embolism or severe bleeding within 6 months before the first administration；
14. Combined symptomatic brain metastasis, meningeal metastasis, spinal cord tumor invasion, and spinal cord compression syndrome；
15. Use of strong inhibitors or inducers of CYP3A, CYP2C8 and UGT1A1 within 14 days before the first administration；
16. Participate in other study and use study drug within 1 month or within 5 half-lives of the drug (whichever comes first) before the first administration；
17. Pregnant or breastfeeding women, or subjects of childbearing age who refuse contraception；
18. Patients who are not suitable to participate in this trial for any reason judged by the investigator；

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2024-06-05 (Estimated); Primary Completion 2025-06-05 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of liposomal irinotecan | 1 months
  Defined as the highest dose of DLT in<33% of subjects .
Objective Response Rate | 5 months
  Defined as the proportion of patients who achieved complete response (CR) and partial response (PR) according to RECIST v1.1.

SECONDARY OUTCOMES:
Dose-Limiting Toxicities (DLT) of liposomal irinotecan | 1 months
  Defined as adverse events that occur during the DLT observation period and are related to the study drug .
Disease Control Rate | 5 months
  Defined as the proportion of patients who achieved complete response (CR), partial response (PR), and stable disease (SD) according to RECIST v1.1.
Duration of Response | 5 months
  Defined as the time from response(when CR or PR is first diagnosed) to disease progression or death due to any cause.
Progression free Survival | 1 years
  Defined as the time between signing the informed consent form to the disease progression (according to RECIST v1.1 criteria) or death due to any cause.
Overall survival | 1 years
  Defined as the time between signing the informed consent form to death due to various causes.

CONTACTS AND LOCATIONS:
Overall Officials: Yanhong Deng, PhD, Principal Investigator — Sixth Affiliated Hospital, Sun Yat-sen University
Locations (1):
- The Sixth Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No